CLINICAL TRIAL: NCT05669664
Title: A Phase 2 Study of Darolutamide in Combination With Leuprolide Acetate in Hormone-Therapy Naive Recurrent and/or Metastatic Androgen Receptor (AR) Positive Salivary Gland Cancer
Brief Title: Testing the Anti-cancer Drug Darolutamide in Patients With Testosterone-Driven Salivary Gland Cancers
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-10701; NCI-2022-10701 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10553 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10553 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2022-12-30; First posted 2023-01-03 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Salivary Gland Carcinoma; Metastatic Salivary Gland Carcinoma; Recurrent Salivary Gland Carcinoma; Unresectable Salivary Gland Carcinoma
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Biopsy; Specimen Handling; darolutamide; Leuprolide; luprolide acetate gel depot; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (darolutamide, leuprolide acetate) (Experimental): Patients receive darolutamide PO BID on days 1-28 of each cycle and leuprolide acetate IM every 4 or 12 weeks. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy, collection of blood samples, and CT/MRI throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Darolutamide; Drug: Leuprolide Acetate; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Darolutamide — Given PO
  Other Names: Antiandrogen ODM-201; BAY 1841788; BAY-1841788; BAY1841788; Nubeqa; ODM 201; ODM-201; ODM201
Drug: Leuprolide Acetate — Given IM
  Other Names: A 43818; A-43818; A43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Fensolvi; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Luprodex Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Lutrate; Procren; Procrin; Prostap; TAP 144; TAP-144; TAP144; Trenantone; Uno-Enantone; Viadur
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI

SUMMARY:
This phase II trial tests how well darolutamide and leuprolide acetate work in treating patients with androgen receptor positive salivary cancer that has spread from where it first started (primary site) to other places in the body (metastatic), cannot be removed by surgery (unresectable) or that has come back after a period of responding to prior therapy (recurrent). Darolutamide is in a class of medications called androgen receptor inhibitors. It works by blocking the effects of androgen (a male reproductive hormone) to stop the growth and spread of cancer cells. Leuprolide acetate is in a class of medications called gonadotropin-releasing hormone (GnRH) agonists. It works by decreasing the amount of certain hormones in the body. Giving darolutamide in combination with leuprolide acetate may help to stop the growth of tumor cells that need androgens to grow or shrink them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the best overall response rate (BOR) of recurrent/metastatic androgen receptor positive (AR+) salivary gland cancer (SGC) patients within one year of darolutamide and androgen deprivation therapy (ADT).

SECONDARY OBJECTIVES:

I. To evaluate progression-free survival (PFS). II. To evaluate overall survival (OS). III. To evaluate toxicity by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.

EXPLORATORY OBJECTIVES:

I. To evaluate molecular, genomic and transcriptomic biomarkers in serial research biopsies obtained before and on darolutamide and ADT.

II. To evaluate the differences in BOR, PFS, OS with darolutamide and ADT treatment among patients who did and did not receive prior systemic therapy for AR+ SGC.

OUTLINE:

Patients receive darolutamide orally (PO) twice daily (BID) on days 1-28 of each cycle and leuprolide acetate intramuscularly (IM) every 4 or 12 weeks. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy, collection of blood samples, and computed tomography (CT)/magnetic resonance imaging (MRI) throughout the trial.

After completion of study treatment, patients are followed every 3-6 months for 2 years after treatment discontinuation or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed salivary gland cancer that is recurrent/metastatic or unresectable/locally advanced, with AR expression detected by immunohistochemistry (IHC) on a Clinical Laboratory Improvement Act (CLIA)-approved assay. Androgen receptor testing by immunohistochemistry (IHC) can be performed locally in a CLIA (Clinical Laboratory Improvement Amendments) certified lab
* Patients must have measurable disease
* Patients must have not had prior AR-targeted therapy, except for AR-targeted therapy administered in the neoadjuvant and/or adjuvant setting and with disease recurrence more than 6 months since treatment completion
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of darolutamide in combination with leuprolide acetate in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (exception: patients with elevated bilirubin due to Gilbert's disease would be eligible for the trial)
* Aspartate aminotransferase (AST) (serum (glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase ([SGPT]) =< 3 x institutional ULN
* Creatinine =< 1.5 x institutional ULN
* Glomerular filtration rate (GFR) >= 30 mL/min/1.73 m^2 (by Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI])
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* The effects of darolutamide on the developing human fetus are unknown. For this reason and because androgen receptor inhibitor agents as well as other therapeutic agents used in this trial are known to be teratogenic (leuprolide-acetate), women of child-bearing potential and men must agree to use adequate contraception (non-hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men and women treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 7 days after completion of darolutamide administration or after the depot interval for the leuprolide-acetate dose used has been completed, whichever is longer
* Ability to understand and the willingness to sign a written informed consent document
* Patients must have tumors that are safely accessible for biopsy.

  * Note: Two research biopsies are mandated in this trial. If the biopsy is deemed to be unsafe after attempting the first biopsy, the patient will remain eligible for the trial and subsequent tumor biopsies will not be required

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia and peripheral neuropathy
* Patients with a vascular or ischemic event within 6 months of study registration
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to darolutamide or leuprolide acetate
* Patients on combined P-gp and strong or moderate CYP3A inducers or BCRP substrates are excluded. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with uncontrolled intercurrent illness
* Pregnant women are excluded from this study because darolutamide is an androgen receptor inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with darolutamide and leuprolide-acetate, breastfeeding should be discontinued if the mother is treated with darolutamide and leuprolide-acetate. These potential risks may also apply to other agents used in this study.
* Patients with moderate hepatic impairment (Child-Pugh Class B or C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2027-04-11 (Estimated); Study Completion 2027-04-11 (Estimated)

PRIMARY OUTCOMES:
Best overall response (BOR) | Within 1 year of initiating treatment
  The trial will be considered positive if 8 or more complete response/partial response are observed in stage 1 and stage 2 combined.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From day 1 of treatment until progression or death, assessed up to 2 years
  Will be estimated using Kaplan-Meier methodology. Patients without an event (progression, death) will be censored at the time of last follow-up or last day known to be alive.
Overall survival (OS) | From day 1 of treatment until progression or death, assessed up to 2 years
  Will be estimated using Kaplan-Meier methodology. Patients without an event (progression, death) will be censored at the time of last follow-up or last day known to be alive.
Incidence of adverse events (AEs) | Up to 2 years
  Will be listed individually per patient according to Common Terminology Criteria for Adverse Events version 5.0, and the number of patients experiencing each AE will be summarized.

OTHER OUTCOMES:
Molecular, genomic, and transcriptomic biomarkers | Up to 2 years
  Will be summarized by descriptive statistics, including mean, median and standard deviation for continuous biomarker data and frequency (%) for categorical data. Differences in a biomarker at baseline, on treatment, and change between those two time points amongst responders and non-responders will be compared using Fisher's exact tests for categorical biomarker data and Wilcoxon Rank-Sum tests for continuous biomarker data. In addition, a Cox proportional hazards model will be used to explore the prognostic relationship for these biomarkers measured at baseline and PFS and OS.
Differences in BOR, PFS, OS in patients who did and did not receive prior systemic therapy for androgen receptor positive salivary gland cancer | Up to 2 years
  The BOR, PFS, and OS with darolutamide plus androgen deprivation therapy in patients with and without prior systemic therapies for recurrent/metastatic/unresectable disease will be compared using Fisher's exact for binary outcome and log-rank test for time-to-events outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Alan L Ho, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (27):
- United States (27):
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Emory University Hospital Midtown, Atlanta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm